CLINICAL TRIAL: NCT01901172
Title: A Study of the Drug-Drug Interaction of RO5503781 and Posaconazole, the Relative Bioavailability of New Formulations of RO5503781 and the Food-Effect on the Pharmacokinetics of RO5503781 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: NP28902
Record Dates: First submitted 2013-07-09; First posted 2013-07-17 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — posaconazole

ARMS (4):
- Extension (Experimental)
  Interventions: Drug: RO5503781
- Part 1: Drug-drug interaction (Experimental)
  Interventions: Drug: RO5503781; Drug: posaconazole
- Part 2: Relative bioavailability (Experimental)
  Interventions: Drug: RO5503781
- Part 3: Food effect (Experimental)
  Interventions: Drug: RO5503781

INTERVENTIONS:
Drug: RO5503781 — Single dose on Day 1 (high fat, low fat, or fasted), Day 10 (fasted, low fat, or high fat), and Day 19 (low fat, fasted, or high fat) in a crossover design
  Arms: Part 3: Food effect
Drug: RO5503781 — Daily for 5 days followed by 23 days rest per cycle
  Arms: Extension
Drug: RO5503781 — Single doses of current formulation, optimized MBP formulation and new SDP formulation, Days 1, 8 and 15 in a crossover design
  Arms: Part 2: Relative bioavailability
Drug: RO5503781 — Single doses Days 1 and 11
  Arms: Part 1: Drug-drug interaction
Drug: posaconazole — Multiple doses Days 8-14
  Arms: Part 1: Drug-drug interaction

SUMMARY:
This multicenter, open-label study will evaluate the effect of posaconazole on the pharmacokinetics of RO5503781, the relative bioavailability of two new RO5503781 formulations, and the effect of food on the pharmacokinetics of RO5503781 in patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Histologically or cytologically confirmed advanced malignancies, except all forms of leukemia and lymphoma, for which standard curative or palliative measures do not exist, are no longer effective, or are not acceptable to the patient
* Measureable or evaluable disease (by RECIST criteria version 1.1 for solid tumors prior to the administration of study drug
* Life expectancy of >/= 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Female patients of childbearing potential and male patients who are not surgically sterile must be willing to use effective methods of contraception as defined by protocol during the treatment period and for 10 days after the last dose of RO5503781.
* There are no limitations on additional, allowable type and amount of prior anti-tumor therapy. Acute toxicities from any prior anti-tumor therapy, surgery, or radiotherapy must have resolved to NCI-CTCAE version 4.03 Grade </= 1. The last dose of prior therapy must >/= 21 days prior to the first administration of study drug RO5503781 (or >/= 5 x terminal half-life of that therapy).
* Adequate bone marrow, hepatic and renal function
* Patients with stable CNS metastases (have had therapy or do not require therapy, are off steroids, have no change on screening CT or MRI and are asymptomatic), are eligible

Exclusion Criteria:

* Any form of leukemia except for Stage 0 and 1 chronic lymphocytic leukemia (CLL) not requiring treatment in addition to the underlying malignancy
* Hormonal therapy within the 2 weeks prior to the first dose of study medication. Patients with prostate cancer who are not surgically castrated should remain on GnRH analogues.
* Patients who are using other investigational agents or who received investigational drugs </= 4 weeks prior to study treatment start.
* Pre-existing GI disorders that may interfere with proper absorption of the drug(s), as per investigator discretion.
* History of allergic reactions attributed to components of the formulated product
* History of seizure disorders or unstable CNS metastases
* Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* Patients who must receive CYP2C8 inhibitors, substrates or inducers, strong CYP 3A4 inducers or moderate/strong CYP3A4 inhibitors listed in protocol while on study. Substrates, inducers, and inhibitors listed in protocol must be discontinued 7 or 14 days prior to start of study medication.
* Evidence of electrolyte imbalance (treatment for correction of electrolyte imbalances is permitted during screening to meet eligibility)
* Pregnant or breast feeding women
* HIV-positive patients who are currently receiving combination anti-retroviral therapy
* Patients with known coagulopathy, platelet disorder or history of non-drug induced thrombocytopenia.
* Patients receiving oral or parenteral anticoagulants/antiplatelet agents (e.g., chronic daily treatment with aspirin (> 325 mg/day), clopidogrel, low molecular weight heparin, or subcutaneous anticoagulant prophylaxis). A washout period of at least 7 days prior to the start of study is required. Patients may receive anticoagulant flushes for maintenance of indwelling catheters.
* Patients who refuse to potentially receive blood products and/or have a hypersensitivity to blood products
* Part 1 only: Hypersensitivity to posaconazole, or any of the other ingredients, or any other azole antifungal
* Part 1 and Part 3: Patients who cannot tolerate high-fat and/or full meals.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Part 1: Area under the concentration-time curve (AUC) | 22 days
Part 1: Maximum concentration (Cmax) | 22 days
Part 1: Change in serum macrophage inhibitory cytokine-1 (MIC-1) | from baseline to Day 22
Part 2: Relative bioavailability: Area under the concentration-time curves (AUCs) | 22 days
Part 3: Food effect: Area under the concentration-time curves (AUCs) | 28 days

SECONDARY OUTCOMES:
Safety: Incidence of adverse events in combination with posaconazole | 28 days
Safety: Incidence of adverse events (new formulations) | 28 days
Safety: Incidence of adverse events (optional treatment extension) | approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- United States (2):
  - Scottsdale, Arizona
  - Dallas, Texas
- Canada (2):
  - Toronto, Ontario
  - Montreal, Quebec